CLINICAL TRIAL: NCT04496349
Title: A Phase IIa Study Evaluating the Pharmacokinetics, Safety and Efficacy of APG-115 as a Single Agent or in Combination With APG-2575 in Subjects With Relapsed/Refractory T-Cell Prolymphocytic Leukemia (R/R T-PLL) or Non-Hodgkin's Lymphoma (NHL).
Brief Title: A Study Evaluating APG-115 as a Single Agent or in Combination With APG-2575 in Subjects With R/R T-PLL and NHL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ascentage Pharma Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APG115TU101
Record Dates: First submitted 2020-07-22; First posted 2020-08-03 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: T-Prolymphocytic Leukemia; Non-Hodgkins Lymphoma
MeSH Terms: conditions — Leukemia, Prolymphocytic, T-Cell; Lymphoma, Non-Hodgkin | interventions — Lisaftoclax

STUDY DESIGN:
Intervention Model Description: The study consists of Part 1 APG-115 as monotherapy. Part 2 APG-2575 in combination with APG-115 dose escalation and APG-2575 in combination with APG-115 dose expansion phase. APG-115 and APG-2575 will be orally administrated on 21-day cycles. Patients will receive APG-115 QOD, 2 weeks on, 1 week off, and APG-2575 QD, in repeated 21-day cycles.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- APG-115 monotherapy part (Experimental): APG-115 will be given alone
  Interventions: Drug: APG-115
- APG-115 + APG-2575 combination dose escalation part (Experimental): APG-115 is given in combination with APG-2575
  Interventions: Drug: APG-115; Drug: APG-2575
- APG-115 + APG-2575 combination dose expansion part (Experimental): APG-115 is given in combination with APG-2575
  Interventions: Drug: APG-115; Drug: APG-2575

INTERVENTIONS:
Drug: APG-115 — QOD, 2 weeks on, 1 week off, in repeated 21-day cycles
Drug: APG-2575 — APG-2575 given orally each day in cycle, in repeated 21-day cycles
  Arms: APG-115 + APG-2575 combination dose escalation part; APG-115 + APG-2575 combination dose expansion part

SUMMARY:
The goal of this study is to evaluate the pharmacokinetics (PK), safety, and efficacy of APG-115 as a single agent or in combination with APG-2575 in patients with T-PLL and NHL.

DETAILED DESCRIPTION:
This is a phase IIa, open-label, multi-center, clinical trial of interfering the binding of MDM2 oncoprotein with the tumor suppressor P53 protein, leads to increased P53 and P21 protein expression and activates P53-mediated apoptosis. The hypothesis is that APG-115 monotherapy and in combination with APG-2575 will shows good safety and efficacy in patients with R/R T-PLL and NHL

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Patients with relapsed/refractory T-PLL who have active disease and have received at least one prior therapy; Patients with histologically confirmed diagnosis of NHL, NHL Patients must be either relapsed, refractory, intolerant, or are considered ineligible for therapies known to provide clinical benefit;
3. Patients must not have had chemotherapy or antibody therapy for 7 days prior to starting APG-115 and/or APG-2575. However, patients with rapidly proliferative disease may receive hydroxyurea or decadron until 24 hours prior to starting therapy on this protocol.
4. Absolute neutrophil count (ANC) ≥ 500/mm˄3; hemoglobin ≥ 60 g/L; platelet count ≥ 30,000/mm˄3
5. Patients with adequate organ function;
6. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2;
7. Patient must have the ability to understand the requirements of the study and signed informed consent. A signed informed consent by the patient or his/her legally authorized representative is required prior to their enrollment on the protocol.

Exclusion Criteria:

1. Patient previously treated with a murine double minute 2 (MDM2) inhibitor.
2. Known active, uncontrolled central nervous system (CNS) malignancy
3. Patients require graft versus host therapy, or require continued treatment with systemic immunosuppressive agents (calcineurin inhibitors within 4 weeks prior to the first dose of study drug).
4. Patients who have any conditions or illness that, according to the opinions of the Investigators or the medical monitor, would compromise patient safety or interfere with the evaluation of safety and efficacy to the study drug(s).
5. Patients who have used strong CYP2C8 inhibitors, or moderate or strong CYP3A4 inhibitors or inducers within washout period of 14 days or 7 half-lives before the first administration of study drugs, whichever is longer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2021-07-12 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose of APG-115 | 21 days
  To evaluate the safety of APG-115 as a single agent
Maximum tolerated dose of APG-115+APG-2575 | 21 days
  To evaluate the maximum tolerated dose of APG-115 and APG-2575 in combination

CONTACTS AND LOCATIONS:
Overall Officials: Yifan Zhai, MD, PhD, Study Chair — Ascentage Pharma Group Inc.
Locations (1):
- MD Anderson, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No